CLINICAL TRIAL: NCT05269212
Title: Objectifying Performance Assessments and Personalized Rehabilitation Trajectories to Improve Return to Work in Patients With Persistent Spinal Pain Syndrome Type II: a Randomized Controlled Trial.
Brief Title: Return to Work for Persistent Spinal Pain Syndrome Type II Patients
Acronym: OPERA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moens Maarten (Other)
Collaborators: Vrije Universiteit Brussel (Other); University Ghent (Other); KU Leuven (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPERA
Record Dates: First submitted 2022-02-08; First posted 2022-03-07 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Failed Back Surgery Syndrome; Spinal Cord Stimulation
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator)
  Interventions: Other: Usual Care trajectory
- Personalized biopsychosocial rehabilitation program (Active Comparator)
  Interventions: Other: A biopsychosocial rehabilitation program

INTERVENTIONS:
Other: Usual Care trajectory — Usual care after Spinal Cord Stimulation implantation
  Arms: Usual care
Other: A biopsychosocial rehabilitation program — A personalized biopsychosocial rehabilitation program specifically targeting return to work.
  Arms: Personalized biopsychosocial rehabilitation program

SUMMARY:
A multicenter randomized controlled trial will be conducted to evaluate whether the ability to work in Persistent Spinal Pain Syndrome Type II (PSPS-T2) patients after SCS implantation is different after a personalized biopsychosocial rehabilitation program specifically targeting return to work (RTW) compared with usual care.

DETAILED DESCRIPTION:
A multicenter randomized controlled trial will be conducted to evaluate whether the ability to work in Persistent Spinal Pain Syndrome Type II patients after SCS implantation is different after a personalized biopsychosocial rehabilitation program specifically targeting return to work compared with usual care.

The primary scientific objective is to examine whether the ability to work in PSPS-T2 patients after SCS implantation is different with a personalized biopsychosocial rehabilitation program specifically targeting RTW, compared to usual care. The secondary objective of the study is to examine if a personalized biopsychosocial rehabilitation program specifically targeting RTW, compared to usual care, is different in improving functional capacity, improving work status and participation, obtaining pain relief, increasing health-related quality of life, increasing functioning and physical activity, improving sleep quality, decreasing kinesiophobia, increasing self-management, decreasing anxiety and depression and decreasing healthcare expenditure.

Patients will be randomly allocated (1:1 ratio) to a personalized rehabilitation program or usual care using random, permuted blocks of 2 or 4 patients stratified by investigational site and the duration of sick leave. Participants randomly allocated to the usual care intervention will undergo the usual care trajectory. This program is delivered at each of the participating centres. Patients will follow the usual care as it is implemented in Belgian hospitals, after SCS implantation. Participants randomly allocated to the personalized biopsychosocial return to work program will receive an individualized 14-week rehabilitation program. Therapy is provided at each implantation centres and will start 6 weeks after definitive SCS implantation. Within a 14-week period, patients in this group receive treatment sessions from trained physiotherapists, occupational therapists and psychologists. All therapists will be trained by experts in the different therapy modalities.

Outcome assessments will take place at baseline, immediately before the intervention, immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Persistent Spinal Pain Syndrome Type II (PSPS-T2)
* Chronic pain as a result of PSPS-T2 that exists for at least 6 months with a pain intensity of at least 4/10 on the Numeric Rating Scale, refractory to conservative treatment.
* Dutch speaking persons
* Patient has been informed of the study procedures and has given written informed consent
* Patient willing to comply with study protocol including attending the study visits

Exclusion Criteria:

* Suffering from another chronic illness characterised by chronic generalized widespread pain (e.g. rheumatoid arthritis, fibromyalgia, chronic fatigue syndrome, scleroderma).
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Work ability | The change between the baseline screening and the evaluation immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.
  Work ability, evaluated with the Work Ability Index

SECONDARY OUTCOMES:
Functional capacity evaluation | The change between the baseline screening and the evaluation immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.
  Functional capacity evaluation will be performed using a shortened version of the Isernhagen Work Systems.
Work status and participation | The change between the baseline screening and the evaluation immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.
  Work Rehabilitation Questionnaire will be used to evaluate functioning in Vocational Rehabilitation
Overall pain intensity with Visual Analogue Scale (VAS) | The change between the baseline screening and the evaluation immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.
  Overall pain, defined as a combination of back and leg pain, but not pain from other body parts, measured with the VAS (100mm).
Health related quality of life | The change between the baseline screening and the evaluation immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.
  Health related quality of life, evaluated with the EuroQol with five dimensions and 5 levels.
Physical activity | The change between the baseline screening and the evaluation immediately after the intervention, 6 months after the intervention and 12 months after the intervention.
  Physical activity will be objectively measured with actigraphy.
Functional disability | The change between the baseline screening and the evaluation immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.
  The functional disabilities will be assessed with the Oswestry Disability Index (ODI).
Sleep quality | The change between the baseline screening and the evaluation immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.
  Perceived sleep quality will be measured with the Pittsburgh Sleep Quality Index.
Kinesiophobia | The change between the baseline screening and the evaluation immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.
  The Tampa Scale for Kinesiophobia will be used to measure kinesiophobia.
Healthcare utilisation | The change in healthcare utilisation starting from the the baseline screening up to 12 months after the intervention.
  Healthcare expenditure will be investigated by self-reporting methods.
Anxiety and depression | The change between the baseline screening and the evaluation immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.
  The hospital Anxiety and Depression Scale (HADS) will measure symptoms of anxiety and depression.
Patients' individual competencies for self-management | The change between the baseline screening and the evaluation immediately after the intervention, 3 months after the intervention, 6 months after the intervention and 12 months after the intervention.
  Patient activation measure-13 (PAM) is a 13-item instrument which assesses self-reported behaviour, knowledge, and confidence for self-management of one's health.

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (5):
  - UZ Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - Universitair Ziekenhuis Brussel, Jette
  - AZ Nikolaas, Sint-Niklaas
  - AZ Turnhout, Turnhout

REFERENCES:
- [Derived] Moens M, Goudman L, Van de Velde D, Godderis L, Putman K, Callens J, Lavreysen O, Ceulemans D, Leysen L; OPERA consortium; De Smedt A. Personalised rehabilitation to improve return to work in patients with persistent spinal pain syndrome type II after spinal cord stimulation implantation: a study protocol for a 12-month randomised controlled trial-the OPERA study. Trials. 2022 Dec 5;23(1):974. doi: 10.1186/s13063-022-06895-5. PMID 36471349